CLINICAL TRIAL: NCT06818617
Title: Analysis of Changes in Blood Glucose Using a Continuous Blood Glucose Monitoring After Spinal Epidural Nerve Block with Steroids in Patients with Low Back Pain
Brief Title: Analysis of Changes in Blood Glucose Spinal Epidural Nerve Block with Steroids in Patients with Low Back Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sung Hyun Lee (Other)
Responsible Party: Sponsor-Investigator, Sung Hyun Lee, Kangbuk Samsung Hospital, Kangbuk Samsung Hospital
Organization: Kangbuk Samsung Hospital (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-12-014
Record Dates: First submitted 2025-02-07; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Glucose Level Change
Keywords: continous glucose monitering

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- dexamethasone dose-0 (Active Comparator)
  Interventions: Procedure: Epidural steroid injection (ESI)
- dexamethasone dose 5.0 (Active Comparator)
  Interventions: Procedure: Epidural steroid injection (ESI)
- dexamethasone dose-7.5 (Active Comparator)
  Interventions: Procedure: Epidural steroid injection (ESI)

INTERVENTIONS:
Procedure: Epidural steroid injection (ESI) — epidural nerve block procedures for patients with spinal conditions such as stenosis or disc herniation

SUMMARY:
This study aims to investigate the effect of different doses of dexamethasone used in epidural nerve block procedures on blood sugar levels. Patients with spinal conditions such as stenosis or disc herniation will be enrolled. Blood glucose and HbA1c levels will be measured before the procedure, and participants will use continuous glucose monitoring devices for 2-3 days before the procedure. They will be randomly assigned to one of three groups: no dexamethasone, 5mg dexamethasone, or 7.5mg dexamethasone. Blood glucose will be monitored for one week after the procedure, and follow-up will be done two weeks later to assess pain and blood sugar data. This study will help determine how steroid doses affect blood sugar, especially in elderly patients, and provide more accurate information than previous studies.

ELIGIBILITY:
Inclusion Criteria:

* patients need to epidural steroid injection for treating back pain
* patients diagnosed with diabetes or prediabetes.

Exclusion Criteria:

* Patients with poorly controlled blood sugar.(HbA1c>8.5)

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-02-19 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Glucose change | glucose change between befor intervention and after for 7days.

IPD SHARING:
Plan to Share IPD: Yes
Format of data(anonymized datasets).
Supporting Information: Study Protocol, SAP
Time Frame: Start date: The date when the individual participant data (IPD) and supporting information will first be made available.( starting the study)
  End date: The date when access to the IPD and supporting information will no longer be available or when the sharing period ends. (for 3yrs)